CLINICAL TRIAL: NCT02873364
Title: High Dose Vitamin D Supplementation in Treatment of Chronic Spontaneous Urticaria
Brief Title: High Dose Vitamin D Supplementation in Chronic Spontaneous Urticaria
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Keramatallah Jahanshahi, Resident of internal medicine, Shiraz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 93-01-01-8312
Record Dates: First submitted 2016-08-11; First posted 2016-08-19 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-08

CONDITIONS: Urticaria
MeSH Terms: conditions — Urticaria | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin D3 (Low dose) (Active Comparator): Daily 600 unites of vitamin D + Cetirizine 10mg twice a day
  Interventions: Drug: Vitamin D3 (Low dose)
- Vitamin D3 (High dose) (Experimental): Daily 4000 unites vitamin D + Cetirizine 10mg twice a day
  Interventions: Drug: Vitamin D3 (High dose)

INTERVENTIONS:
Drug: Vitamin D3 (High dose) — Daily 4000 unites vitamin D
  Other Names: cholecalciferol
  Arms: Vitamin D3 (High dose)
Drug: Vitamin D3 (Low dose) — Daily 600 unites vitamin D
  Other Names: cholecalciferol
  Arms: Vitamin D3 (Low dose)

SUMMARY:
Chronic spontaneous urticaria is an inflammatory disease which is characterized with intermittent or daily urticaria. This diseases lasts for more than 6 weeks. Several recent studies have suggested a role for vitamin D in modulation of immune system and pathogenesis of chronic urticaria.

ELIGIBILITY:
Inclusion Criteria:

* Uriticaria or angioedema daily or more than 3 days a weeks for at least 6 weeks

Exclusion Criteria:

* Physical urticaria aquired or hereditary angioedema Calcium level > 10.3 mg/dl Glomerular filtration rate <50 Sarcoidosis Primary hyperparathyroidism Granulomatous diseases Malignancies Pregnancy Lactation

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-08; Primary Completion 2016-12 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Urticaria symptom severity questionnaire after 1 week | 1 weeks
  Urticaria Symptom Severity ranging from 0 to 93

SECONDARY OUTCOMES:
Urticaria symptom severity questionnaire after 6 week | 6 weeks
  Urticaria Symptom Severity ranging from 0 to 93
Urticaria symptom severity questionnaire after 12 week | 12 weeks
  Urticaria Symptom Severity ranging from 0 to 93

CONTACTS AND LOCATIONS:
Overall Officials: Keramatallah Jahanshahi, MD, Principal Investigator — Shiraz University of Medical Sciences
Locations (1):
- Shiraz University of Medical Sciences, Shiraz, Fars, Iran

IPD SHARING:
Plan to Share IPD: Yes